CLINICAL TRIAL: NCT04015219
Title: A Prospective, Randomized, and Controlled Clinical Study to Evaluate PROKERA® in the Management of Signs and Symptoms Associated With Dry Eye Disease
Brief Title: Management of Signs and Symptoms Associated With Dry Eye Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment constraints
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROKERA-CS001
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment Arm (Experimental): PROKERA SLIM + Standard of Care
  Interventions: Device: Self retained cryopreserved amniotic membrane; Other: lifitegrast ophthalmic solution
- Control Arm (Active Comparator): Standard of Care
  Interventions: Other: lifitegrast ophthalmic solution

INTERVENTIONS:
Device: Self retained cryopreserved amniotic membrane — PROKERA SLIM
  Arms: Treatment Arm
Other: lifitegrast ophthalmic solution — Xiidra® (5% lifitegrast ophthalmic solution, Shire, Lexington, MA)
  Other Names: Xiidra

SUMMARY:
A prospective randomized, and controlled study to compare the effectiveness of PROKERA® SLIM plus standard of care (SOC) in the PROKERA® SLIM Arm to SOC alone in the Control Arm. Subjects presenting with moderate DED defined as corneal fluorescein staining score of ≥ 3 points out of 9 will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate dry eye defined as corneal fluorescein staining score of ≥ 3
* Age ≥ 18 years
* Distance best corrected visual acuity better than 20/60 Snellen equivalent in each eye
* Willing to sign a written informed consent to participate
* Able to follow study instructions, with the intention of completing all required visits

Exclusion Criteria:

* Presence of persistent corneal epithelial defect or ulcer in either eye
* Presence of active ocular infection in either eye
* Presence of ocular inflammation that is not related to keratoconjunctivitis sicca, e.g., allergy, severe blepharitis
* Presence of other corneal disorder(s) that give rise to reduced corneal sensitivity, such as recurrent herpes keratitis
* Presence of corneal diseases other than dry eye that can disturb the pre-corneal tear film such as epithelial basement membrane dystrophy (EBMD)
* Contact lens wear
* History of recent ocular surgery/trauma, which could affect corneal sensitivity, e.g., corneal transplantation, LASIK
* Presence of cicatricial ocular surface diseases
* A medical or ocular condition, or a personal situation, which in the principal investigator's opinion, is not appropriate for participation in the trial
* Any scheduled or planned ocular or systemic surgery or procedure during the study
* Pregnancy and women who are expecting to be pregnant.
* Current enrolment in another interventional drug or device study or participation in such a study within 30 days of anticipated entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Excellence in Eye Care, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: PROKERA SLIM + Standard of Care
  PROKERA SLIM is a self retained cryopreserved amniotic membrane that is inserted once for 5 ±1 days
Period: Overall Study
Arm/Group | Treatment Arm | Control Arm
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control Arm | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (4.2) | 46 (0) | 63 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Corneal Fluorescein Staining
Description: corneal fluorescein staining score of study eye graded from 0 to 9, with a score of 9 being worse. The corneal fluorescein staining score is the sum of three scores by subdividing the entire cornea into upper 1/3, middle 1/3, and lower 1/3, of which each is graded from 0 (no staining) to 3 (diffuse staining).
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 2 | 1
units on a scale | 0.5 (0.7) | 3 (0)

2. Secondary Outcome: Eye Dryness Score
Description: Patient subjectively evaluates eye dryness score using a visual analog scale from 0 to 100 maximal discomfort
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 2 | 1
units on a scale | 57.5 (46) | 75 (0)

3. Secondary Outcome: Ocular Surface Disease Index (OSDI)
Description: Patient subjectively evaluates OSDI questionnaire, OSDI is scored on a scale of 0 to 100, with higher scores representing greater disability
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 2 | 1
units on a scale | 64.5 (35) | 52 (0)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Treatment Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT04015219/Prot_SAP_000.pdf